CLINICAL TRIAL: NCT04291872
Title: Randomized Clinical Trial of Heated High-Viscosity Glass Ionomer Class II Restorations in Primary Molars: 12 Months Follow Up
Brief Title: Heated Glass Ionomer Cement in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarmaraU
Record Dates: First submitted 2020-02-17; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries; Glass-Ionomer Cement; Primary Teeth
MeSH Terms: conditions — Dental Caries | interventions — Glass Ionomer Cements

STUDY DESIGN:
Intervention Model Description: Randomised Control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Heated Arm (Experimental): Proximal cavities were restored with Equia Forte (GC Corporation, Europe) according to manufacturer's orders.
  Interventions: Other: Glass -Ionomer Cement with /without Led Light Cure
- Heated Arm (Experimental): Teeth were restored as same protocole with non-Heated Group. LED light (GC- D-Light DUO) was used at standard mode 1200 mW/cm2, at 50-60 ºC, for 60 sec.
  Interventions: Other: Glass -Ionomer Cement with /without Led Light Cure

INTERVENTIONS:
Other: Glass -Ionomer Cement with /without Led Light Cure — Teeth were restored as same protocole with non-Heated Group. LED light (GC- D-Light DUO) was used at standard mode 1200 mW/cm2, at 50-60 ºC, for 60 sec.

SUMMARY:
Objective: The aim of this study was to assess the influence of heated in the clinical success of proximal high viscosity glass ionomer cement (GIC) restorations in primary molars.

Material & Method: This randomized, split mouth, multicenter study was performed in four different centers including 88 patients aged between 5-7 years old. Selection criteria included clinically and/or radiographically detected proximal caries extending into the dentin tissue. A total of 250 primary molars were restored with a bulk fill GIC (Equia Forte, GC, Europe) and randomly allocated to one of the following groups: 1) non-heated (n = 125) and 2) heated (n = 125). LED light (GC- D-Light DUO, Tokyo Japan) was used at standard mode 1200 mW/cm2, at 50-60 ºC, for 60 sec for heat application. All restorations were clinically evaluated using modified USPHS criteria at the baseline, 6 months and 12 months. Chi-square test, Fisher's Exact Chi-square test, Continuity (Yates) correction, Fisher Freeman Halton test and Mc Nemar test were used to compare qualitative data with descriptive statistical methods (frequency). Kaplan Meier and Life Tables were used for survival analysis. P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is mentally and systemically healthy
* Subject has at least two approximal carious lesions at both sides of jaws
* Subject has a normal occlusal relationship with natural dentition
* Subject has at least one adjacent tooth contact

Exclusion Criteria:

* Subject has history of bruxism,
* Subject has allergies to ingredients of glass ionomer based restorative materials.
* Cavity/Caries has highly mineralized pigmented lesions, hypoplasia, fracture or cracks,
* Subject has abrasion, erosion, abfraction,
* Subject has fistula, abscess or pathological mobility,
* Subject has pain, pulp exposure

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Clinical success assessment measurement | 12 months.
  All restorations were evaluated by using Modified US Public Health Service criteria (modified USPHS criteria). Marginal Integrity (MI)), Marginal Discoloration (MD), Secondary Caries (SC), Anatomic Form (AF), and retention (R) were evaluated. A restoration was considered a failure when codes Charlie (C) and D (Delta) were registered. Codes A (Alpha) and B (Bravo) was considered a success or acceptable. follow up period was baseline, 6th months, 12th months.